CLINICAL TRIAL: NCT04907838
Title: Insulin Stimulated Vasodilation in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Stefan Mortensen, Professor, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: s-20180040
Record Dates: First submitted 2019-05-04; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — cyclo(Trp-Asp-Pro-Val-Leu); BQ 788

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetics (Experimental): BQ123 (25 nmol/min), BQ788 (25 nmol/min)
  Interventions: Drug: Insulin clamp; Drug: BQ123; Drug: BQ123 + BQ788
- Healthy controls (Experimental): BQ123 (25 nmol/min), BQ788 (25 nmol/min)
  Interventions: Drug: Insulin clamp; Drug: BQ123; Drug: BQ123 + BQ788

INTERVENTIONS:
Drug: Insulin clamp — Continous infusion insulin + glucose
Drug: BQ123 — Continuous infusion of Insulin + glucose + BQ123
Drug: BQ123 + BQ788 — Continous infusion of insulin + glucose + BQ123 + BQ788

SUMMARY:
This study evaluates the role of endothelin in insulin stimulated vasodilation and glucose uptake. The subjects will complete an hyperinsulinemic euglycemic clamp with and without blockade of the endothelin receptors.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes OR healthy control (no type 2 diabetes)
* BMI<32

Exclusion Criteria:

* heart disease
* pregnancy or birth within 3 month
* smoking
* Kidney disease
* beta-blockers
* insulin treatment (for type 2 diabetics)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Glucose infusion rate | 3.5 hours
  Glucose infusion rate required to maintain euglycemia during insulin clamp with and without endothelin blockade
Leg blood flow | 3.5 hours
  Effect of endothelin receptor blockade on leg blood flow (ultrasound Doppler) during insulin clamp with and without endothelin blockade

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Mortensen, DMSc, Principal Investigator — Professor
Locations (1):
- Cardiovascular and Renal Research, Odense, Denmark

REFERENCES:
- [Derived] Young BE, Padilla J, Finsen SH, Fadel PJ, Mortensen SP. Role of Endothelin-1 Receptors in Limiting Leg Blood Flow and Glucose Uptake During Hyperinsulinemia in Type 2 Diabetes. Endocrinology. 2022 Mar 1;163(3):bqac008. doi: 10.1210/endocr/bqac008. PMID 35084435